CLINICAL TRIAL: NCT07250776
Title: Effects of Body Awareness Therapy on Physical Psychosocial Outcomes in Peripheral Artery Disease: A Randomized Controlled Trial
Brief Title: Effects of Body Awareness Therapy on Functional Capacity, With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Emre Şenocak, Assistant Professor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/68
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Peripheral Arterial Disease
Keywords: Body Awareness Therapy; rehabilitation
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Body Awareness Therapy Group (Experimental): Physiotherapy and body awareness therapy were applied
  Interventions: Procedure: Body Awareness Therapy; Procedure: Conventional Physiotherapy
- Conventional Therapy Group (Active Comparator): Physiotherapy was applied.
  Interventions: Procedure: Conventional Physiotherapy

INTERVENTIONS:
Procedure: Body Awareness Therapy — The Body Awareness Therapy content included relaxation exercises, breathing exercises, floor exercises for trunk and pelvic movements, and extremity movements. Body Awareness Therapy was also administered 1 x 7 x 8 hours/day/week.
  Arms: Body Awareness Therapy Group
Procedure: Conventional Physiotherapy — The conventional physiotherapy program included breathing and aerobic exercises, energy conservation techniques, and activities of daily living. The exercises were supervised once a week and unsupervised for six days. The program was administered 1 x 7 x 8 hours/day/week.

SUMMARY:
Patients will be divided into two groups. One group will receive only a conventional physiotherapy program. The conventional physiotherapy program included breathing and aerobic exercises, energy conservation techniques, and activities of daily living. The exercises were supervised once a week and unsupervised for six days. The program was administered 1 x 7 x 8 hours/day/week.

The experimental group received Body Awareness therapy in addition to the conventional physiotherapy program. The exercise content included relaxation exercises, breathing exercises, floor exercises for trunk and pelvic movements, and extremity movements. Body Awareness Therapy was also administered 1 x 7 x 8 hours/day/week.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Peripheral Artery Disease (PAD) (confirmed by Doppler ultrasonography or Ankle-Brachial Index (ABI) ≤ 0.90).
* Being between 40 and 75 years of age.
* Having Stage II-III PAD.
* Being able to walk independently or with minimal support.
* Being fit for exercise with cardiac or pulmonary functions.
* Having a cognitive level sufficient to participate in body awareness training.
* Having a stable cardiovascular status (not having had an acute cardiac event, myocardial infarction, or stroke) within the last 6 months.
* Agreeing to actively participate in the study and signing the informed consent form.

Exclusion Criteria:

* Having Stage IV PAD.
* Individuals unable to carry out daily activities due to severe rest pain.
* Serious cardiovascular, pulmonary, neurological, cognitive, or musculoskeletal diseases
* Those who have had a myocardial infarction, stroke, or surgery within the last 6 months.
* Uncontrolled hypertension, heart failure, respiratory failure, or dependence on oxygen support
* Active infection or inflammatory diseases
* Uncontrolled diabetes or renal failure
* Missed 2 consecutive sessions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
6-Minute Walk Test | Baseline
6-Minute Walk Test | End of the 8th week
Muscle Strength | Baseline
  For Quadriceps and Hamstring muscles with hand-held dynamometer
Muscle Strength | End of the 8th week
  For Quadriceps and Hamstring muscles with hand-held dynamometer
Body Awareness Questionnaire (BAQ) | Baseline
  The total score on the scale is between 18 and 126. A high score indicates a high level of awareness.
Body Awareness Questionnaire (BAQ) | End of the 8th week
  The total score on the scale is between 18 and 126. A high score indicates a high level of awareness.
Visual Analog Scale | Baseline
  Durnig resting, at Night and After Training. A high score indicates a high level of pain intensity.
Visual Analog Scale | End of the 8th week
  Durnig resting, at Night and After Training. A high score indicates a high level of pain intensity.
Claudication Onset Distance | Baseline
Claudication Onset Distance | End of the 8th week
Absolute Claudication Distance | Baseline
Absolute Claudication Distance | End of the 8th week
Pain Catastrophizing Scale | Baseline
  The total score ranges from 0 to 52. Higher scores indicate greater levels of pain catastrophizing.
Pain Catastrophizing Scale | End of the 8th week
  The total score ranges from 0 to 52. Higher scores indicate greater levels of pain catastrophizing.
Pittsburgh Sleep Quality Index | Baseline
  The total score ranges from 0 to 21. Higher scores reflect poorer sleep quality.
Pittsburgh Sleep Quality Index | End of the 8th week
  The total score ranges from 0 to 21. Higher scores reflect poorer sleep quality.
Multidimensional Scale of Perceived Social Support | Baseline
  The total score ranges from 12 to 84. Higher scores indicate greater perceived social support.
Multidimensional Scale of Perceived Social Support | End of the 8th week
  The total score ranges from 12 to 84. Higher scores indicate greater perceived social support.
Perceived Stress Scale (PSS-10) | Baseline
  The total score ranges from 0 to 40. Higher scores indicate higher perceived stress.
Perceived Stress Scale (PSS-10) | End of the 8th week
  The total score ranges from 0 to 40. Higher scores indicate higher perceived stress.
Hospital Anxiety and Depression Scale | Baseline
  Each subscale (Anxiety and Depression) ranges from 0 to 21. Higher scores indicate greater anxiety or depressive symptoms.
Hospital Anxiety and Depression Scale | End of the 8th week
  Each subscale (Anxiety and Depression) ranges from 0 to 21. Higher scores indicate greater anxiety or depressive symptoms.
Tampa Scale of Kinesiophobia | Baseline
  The total score ranges from 17 to 68. Higher scores indicate greater fear of movement.
Tampa Scale of Kinesiophobia | End of the 8th week
  The total score ranges from 17 to 68. Higher scores indicate greater fear of movement.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Farabi Hospital, Trabzon, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No